CLINICAL TRIAL: NCT01029015
Title: A Pilot, Phase 4, Sleep Laboratory Study Comparing the Physiology of Nocturnal Bladder Function in Subjects With Overactive Bladder - Associated Nocturia to Subjects With Primary Insomnia and Healthy Normal Subjects
Brief Title: Pilot Trial in Sleep Laboratory Setting to Compare the Physiology of Night Time Bladder Function in Subjects With Overactive Bladder (OAB) Versus Subjects That Have Insomnia and Healthy Normal Subjects
Acronym: Nocturia Plt 1
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sr Manager Clinical Trials Registry, Astellas Pharma Global Development
Other Study IDs: 905-UC-009
Record Dates: First submitted 2009-11-30; First posted 2009-12-09 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2009-11

CONDITIONS: Bladder Function
Keywords: OAB; Insomnia; Bladder function; cystometry; polysomnography
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1 -OAB: Subjects with overactive bladder (OAB)
  Interventions: Procedure: cystometry; Procedure: polysomnography
- Group 2 - Insomnia: Subjects with insomnia
  Interventions: Procedure: cystometry; Procedure: polysomnography
- Group 3 - Normal: Normal Subjects
  Interventions: Procedure: cystometry; Procedure: polysomnography

INTERVENTIONS:
Procedure: cystometry — recording device measuring pressures though catheters placed in bladder and rectum
Procedure: polysomnography — recording device measuring sleep activity through electrodes attached to the subject

SUMMARY:
This is an observational, physiology pilot study of subjects with overactive bladder, insomnia and normal subjects. No study drug will be given. All subjects will complete a one week sleep diary and a 3-day bladder diary. After one week, subjects meeting eligibility requirements will complete a single sleep night stay in a sleep laboratory setting. During the sleep night stay, subjects will be evaluated using cystometry and polysomnography. In the morning following the sleep night stay, subjects will complete a sleep questionnaire and this will complete their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Must not have a urinary tract infection
* Time in bed between 6.5 and 9 hours for at least 5 nights per week for preceding month
* Usual bed time is before midnight (24:00 hours) and typically does not vary by ± 1 hour for preceding month
* OAB subjects

  * OAB symptoms for >= 3 months
  * Documented detrusor overactivity episodes within 6 months
* Insomnia subjects

  * Diagnosis of chronic primary insomnia
  * History of > 1 month of waking up more than 2 times per night and being awake for more than 60 minutes per night for at least 3 months

Exclusion Criteria:

* Diagnosis of both OAB and primary insomnia
* Diagnosis of nocturnal polyuria
* Diagnosis of BPH
* BMI >= 34

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects identified through urology physicians, sleep laboratory physicians and advertising
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2006-11; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Number and proportion of voids associated with urgency | During night in sleep lab
Number and proportion of voids associated with Detrusor Overactivity episodes within 10 minutes prior to the polysomnography (PSG) awakenings | During night in sleep lab
Time from PSG awakening to each void in minutes | During night in sleep lab

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Principal Investigator — Duke University
Locations (1):
- Durham, North Carolina, United States